CLINICAL TRIAL: NCT03153709
Title: A Prospective Cohort Evaluating the Pregnancy Rates and Pharmacokinetic Interactions Among HIV-infected Malawian Women on Efavirenz Initiating the Levonorgestrel Implant or the Depot Medroxyprogesterone Acetate Injectable
Brief Title: Prospective Cohort Evaluating Pregnancy Rates, PK Interactions Among HIV+ Women on EFV Initiating LNG Implant or DMPA
Acronym: FP-ART
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-0471; 1R01HD088279-01A1 (NIH); UNCPM-21701 (Other: UNC)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: HIV Infections
Keywords: Pregnancy rates; pharmacokinetic interactions; Women on efavirenz; initiating the Levonorgestrel Implant; initiating the Depot Medroxyprogesterone Acetate Injectable
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare the pregnancy rates among women who are using the HIV drug Efavirenz and either the birth control injection or implant.

DETAILED DESCRIPTION:
Objective 1: To compare the typical-use pregnancy rates of 710 HIV+ DMPA-users on EFV with 710 HIV+ LNG implant users on EFV through a prospective observational cohort.

The investigators will enroll 710 HIV-infected women on EFV who are initiating the LNG implant and 710 HIV-infected women on EFV who are initiating the DMPA injectable and follow them 1 month after contraceptive initiation and then every 6 months until the end of the 4-year study time period. The investigators will recruit and enroll over a period of 2 years; those who are enrolled at the beginning of the enrollment period may complete up to 4 years of follow-up, whereas those who are enrolled at the end of the 2-year enrollment period will complete 2 years of follow-up. Women will have urine, blood, and hair specimens obtained at each study visit. The primary outcome will be incident pregnancy, evaluated by urine pregnancy testing. The secondary outcome will be contraceptive continuation, evaluated by palpation (for LNG implant) and review of the woman's medical record and study forms (for DMPA). A marginal structural Poisson model will be used to estimate the effect of implant compared to DMPA upon pregnancy incidence. The investigators will adjust for key potential confounders, including frequency of intercourse, age, and body mass index (BMI).

Objective 2: To assess whether greater EFV exposure (measured by hair concentrations) is associated with contraceptive failure in LNG implant users in a 2:1 nested case-control study of 240 LNG implant users.

The investigators estimate that a maximum of 120 pregnancies will occur among LNG implant users in the cohort in Objective 1. From this cohort, the investigators will compare 80 pregnant women who were using the LNG implant at the time of conception and 160 controls who had intercourse during the previous 3 months and were not pregnant after a similar period of LNG implant use. A conditional logistic regression model will be used to assess the association between EFV hair concentrations and contraceptive failure; key potential confounders the investigators will adjust for in the analysis include frequency of intercourse, age, weight, and length of time on EFV. The data for this Objective's exposure, outcome, and confounders will be derived from the Data Collection Forms and study specimens obtained in Objective 1.

Objective 3: To evaluate the effect of EFV 400 mg daily on LNG concentrations among a subset of 25 women enrolled in the prospective cohort study who initiated the LNG implant.

The investigators plan to enroll 25 of the 710 EFV users from their prospective cohort in Objective 1 who are initiating the LNG implant into the pharmacokinetic sub-study. All 25 of these women will be enrolled from 1 health facility, Area 18 Health Centre, and all women will be taking EFV 400 mg daily, which is the standard dose that Malawi will be implementing this year due to its equivalent efficacy but decreased cost and side effects when compared to EFV 600 mg daily. Follow-up visits for women in the sub-study will be conducted at 4, 12, 24, 36, and 48 weeks post-implant initiation. Since these women would already be attending visits at 4, 24, and 48 weeks post-implant initiation, there will only be 2 extra study visits for these sub-study participants at 12 weeks post-implant initiation (Visit 1a) and 36 weeks post-implant initiation (Visit 2a). During the extra Visits 1a and 2a, urine, blood, and hair specimens will be obtained so that pregnancy testing can be performed and blood and hair can be stored for VL, EFV, and LNG testing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years
2. Documented HIV-infected status
3. Current use of EFV
4. Fluency in English or Chichewa (the most commonly-spoken language in Malawi)
5. Not currently pregnant (to be confirmed by urine pregnancy test)
6. Initiation of DMPA or the LNG implant within the past 28 days (to be confirmed by verification in the woman's Health Passport and palpation of the implant if applicable)
7. No use of their current contraceptive during the 3 months before they recently initiated it (i.e., they must be newly starting and not just continuing their chosen contraceptive)
8. No desire for pregnancy in the next 4 years
9. Most recent HIV VL <1,000 copies/mL (as per Malawi guidelines, women who have VL ≥1,000 copies/mL will need to be referred for possible 2nd-line ART without EFV)

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 710 HIV-infected women on EFV who are initiating the LNG implant and 710 HIV-infected women on EFV who are initiating the DMPA injectable
Sampling Method: Non-Probability Sample
Enrollment: 1382 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
pregnancy rates of 710 HIV+ DMPA-users on EFV | 4 years
  urine pregnancy testing
pregnancy rates of 710 HIV+ LNG implant users on EFV | 4 years
  urine pregnancy testing
EFV concentration from blood | 4 years
  A validated HPLC-UV assay for EFV will be used for plasma analysis. Concentrations of EFV in a range of 10 to 10,000 ng/mL will be analyzed.
EFV concentration from hair | 4 years
  Using an IR-MALDESI imaging source coupled to a Thermo Q-Exactive/H-ESI II Bundle mass spectrometer, ~1 cm samples of hair, which will give resultant band intensities over the hair will be analyzed. EFV concentrations at each band intensity will be quantified based on a standard curve.64 Both the total and average concentrations over the 6-month period will be analyzed.
The LNG concentrations from serum | 4 years
  The sensitivity of the LNG is 0.05 ng/ml, and the intraassay and interassay coefficients of variation (CVs) are 4.4% and 8.9%.
HIV viral load from plasma | 4 years
  HIV RNA in the range of 40-10,000,000 copies/mL
DNA quantitated from whole blood | 4 years
  Using a Qiagen DNA extraction kit for blood, 1uL of whole blood will be processed to obtain DNA. This DNA will be quantitated and 120ng will be used in the assay.

SECONDARY OUTCOMES:
contraceptive continuation | 4 years
  palpation (for LNG implant) and review of the woman's medical record and study forms (for DMPA).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tang, MD, MSRC, Principal Investigator — UNC-CH
Locations (1):
- UNC Project, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No